CLINICAL TRIAL: NCT05347043
Title: Evaluation of the Montreal Cognitive Assessment Test as a Screening Tool for Cognitive Dysfunction in in Adults With Sickle Cell Disease
Brief Title: The Montreal Cognitive Assessment.Test in Adults With Sickle Cell Disease
Acronym: EvaCAD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: APHP201174; IDRCB 2021-A01842-39 (Other: ANSM)
Record Dates: First submitted 2022-04-20; First posted 2022-04-26 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Sickle Cell Anemia
Keywords: Sickle cell anemia; cognitive dysfunction; sensitivity and specificity; Diagnostic Techniques and Procedures; Neuropsychological Tests; Montreal cognitive assessment
MeSH Terms: conditions — Anemia, Sickle Cell; Cognitive Dysfunction; Hypersensitivity | interventions — Mental Status and Dementia Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): All patients will undergo both the MoCA test and the standardized neuropsychological evaluation Montreal cognitive assessment and standardized neuropsychological evaluation (Test of Attentional Performance of Zimmermann and Fimm ; Wechsler Adult Intelligence Scale 4th version digit span ; Wechsler memory scale III, spatial span ; Wisconsin Card Scoring Test, GREFEX version ; Wechsler Adult Intelligence Scale 4th version block design ; Six elements test GREFEX version; free and cued selective reminding test, 16 items, B version ; Behavioral Rating Inventory of Executive Function ; Modified Fatigue Impact Scale)
  Interventions: Other: Montreal cognitive assessment

INTERVENTIONS:
Other: Montreal cognitive assessment — Montreal cognitive assessment and standardized neuropsychological evaluation (Test of Attentional Performance of Zimmermann and Fimm ; Wechsler Adult Intelligence Scale 4th version digit span ; Wechsler memory scale III, spatial span ; Wisconsin Card Scoring Test, GREFEX version ; Wechsler Adult Intelligence Scale 4th version block design ; Six elements test GREFEX version; free and cued selective reminding test, 16 items, B version ; Behavioral Rating Inventory of Executive Function ; Modified Fatigue Impact Scale)

SUMMARY:
This study will assess the performances of the Montreal Cognitive Assessment (MoCA) to screen for cognitive impairment in adults with sickle cell anemia. The results of the MoCA and its subscores will be compared to a standardized neuropsychological evaluation using validated tests.

DETAILED DESCRIPTION:
Sickle cell anemia is a monogenic disease affecting the beta-chain of hemoglobin. Cognitive impairment is more prevalent in patients with sickle cell disease than in matched unaffected individuals. Validated tests to screen for cognitive impairment are lacking in this population. Our goal is therefore to assess the performance of the Montreal Cognitive Assessment (MoCA) as a screening tool for cognitive impairment in adults with sickle cell anemia. The results of the MoCA and its subscales will be compared to a standardized neuropsychological evaluation using validated tests.

ELIGIBILITY:
Inclusion Criteria:

* Sickle cell disease, SS or SBêta0 subtypes only
* Attending a consultation or a daycare hospitalization in the Tenon hospital sickle cell center
* Aged 18 years old or more
* Providing written informed consent
* With Health Insurance

Exclusion Criteria:

* Obvious cognitive impairment of neurologic (e.g. previous stroke) or psychiatric origin (e.g. psychotic disorder with negative symptoms)
* Insufficient French language fluency to understand the tests, inability to read and write or with no schooling beyond primary school
* Anticipated unavailability in the next 6 months
* Patients under supervision & guardianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2022-10-20 (Actual); Primary Completion 2024-04-11 (Actual); Study Completion 2024-10-14 (Actual)

PRIMARY OUTCOMES:
sensitivity of a Montreal Cognitive Assessment score < 26 to detect cognitive impairment confirmed by a neuropsychological standardized evaluation | Month 3
  sensitivity of a Montreal Cognitive Assessment score < 26 to detect cognitive impairment defined as an abnormal result in at least one of the following tests : Test of Attentional Performance of Zimmermann and and Fimm (< 5th percentile in at least one of the subscales) ; Wechsler Adult Intelligence Scale 4th version digit span (standard score ≤ 5) ; Wechsler memory scale III, spatial span (standard score ≤ 5) ; Wisconsin Card Scoring Test, GREFEX version (number of categories ≤ 5th percentile or if the number of perseverations is ≥ 95th percentile) Wechsler Adult Intelligence Scale 4th version block design (standard score ≤ 5) ; Six elements test GREFEX version (rank score ≤ 5th percentile ); free and cued selective reminding test, 16 items, B version (Z-score ≤ -1,65 in at least one of the subscales)

SECONDARY OUTCOMES:
specificity of a Montreal Cognitive Assessment score < 26 to detect cognitive impairment confirmed by a neuropsychological standardized evaluation | Month 3
  specificity of a Montreal Cognitive Assessment score < 26 to detect cognitive impairment defined as an abnormal result in at least one of the following tests : Test of Attentional Performance of Zimmermann and Fimm (< 5th percentile in at least one of the subscales) ; Wechsler Adult Intelligence Scale 4th version digit span (standard score ≤ 5) ; Wechsler memory scale III, spatial span (standard score ≤ 5) ; Wisconsin Card Scoring Test, GREFEX version (number of categories ≤ 5th percentile or if the number of perseverations is ≥ 95th percentile); Wechsler Adult Intelligence Scale 4th version block design (standard score ≤ 5) ; Six elements test GREFEX version (rank score ≤ 5th percentile); free and cued selective reminding test, 16 items, B version (Z-score ≤ -1,65 in at least one of the subscales)
sensitivity of a Montreal Cognitive Assessment score < 23 to detect cognitive impairment confirmed by a neuropsychological standardized evaluation | Month 3
  sensitivity of a Montreal Cognitive Assessment score < 23 to detect cognitive impairment defined as an abnormal result in at least one of the following tests : Test of Attentional Performance of Zimmermann and Fimm (< 5th percentile in at least one of the subscales) ; Wechsler Adult Intelligence Scale 4th version digit span (standard score ≤ 5) ; Wechsler memory scale III, spatial span (standard score ≤ 5) ; Wisconsin Card Scoring Test, GREFEX version (number of categories ≤ 5th percentile or if the number of perseverations is ≥ 95th percentile)
  * Wechsler Adult Intelligence Scale 4th version block design (standard score ≤ 5) ; Six elements test GREFEX version (rank score ≤ 5th percentile) ; free and cued selective reminding test, 16 items, B version (Z-score ≤ -1,65 in at least one of the subscales)
sensitivity and specificity of a score ≤ 5/6 in the attention subscale of the Montreal Cognitive Assessment to detect attentional impairment confirmed by a neuropsychological standardized evaluation | Month 3
  sensitivity and specificity of a score ≤ 5/6 in the attention subscale of the Montreal Cognitive Assessment to detect attentional impairment as defined by a Test of Attentional Performance of Zimmermann and Fimm < 5th percentile in at least one of the subscales of the test
sensitivity and specificity of a score ≤ 4/5 in the visuospatial/executive subscale of the Montreal Cognitive Assessment to detect executive impairment confirmed by a neuropsychological standardized evaluation | Month 3
  sensitivity and specificity of a score ≤ 4/5 in the visuospatial/executive subscale of the Montreal Cognitive Assessment to detect executive impairment as defined by an abnormal result in one of the following test : Wisconsin Card Scoring Test, GREFEX version (number of categories ≤ 5th percentile or if the number of perseverations is ≥ 95th percentile); Wechsler Adult Intelligence Scale 4th version block design (standard score ≤ 5) ; Six elements test GREFEX version (rank score ≤ 5th percentile )
sensitivity and specificity of a score ≤ 4/5 in the delayed recall subscale of the Montreal Cognitive Assessment to detect a long term memory impairment confirmed by a neuropsychological standardized evaluation | Month 3
  sensitivity and specificity of a score ≤ 4/5 in the attention subscale of the Montreal Cognitive Assessment to detect attentional impairment as defined by a free and cued selective reminding test, 16 items, B version Z-score ≤ -1,65 (in at least one of the subscales)

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Simon RECH, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Internal Medicine Department - Tenon, Paris, France

IPD SHARING:
Plan to Share IPD: No